CLINICAL TRIAL: NCT01417494
Title: Evaluation of Bevacizumab Combined With First Line Chemotherapy in Patients Aged 75 and Over Suffering From Metastatic Colorectal Adenocarcinoma. Phase II Randomized - Intergroup Trial: FFCD, FNCLCC, GERICO
Brief Title: 1st Line Chemotherapy Alone or With Bevacizumab in Treating Older Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000706869; FFCD-PRODIGE-20 (Other: FFCD); EU-21120 (Other: FFCD); 2010-022080-34 (EudraCT Number)
Record Dates: First submitted 2011-08-13; First posted 2011-08-16 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage IVA colon cancer; stage IVB colon cancer; adenocarcinoma of the rectum; stage IVA rectal cancer; stage IVB rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Drug Therapy; Folfox protocol; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy associated with bevacizumab (Experimental): Chemotherapy (FOLFIRI, FOLFOX, LV5FU2) associated with bevacizumab
  Interventions: Drug: Chemotherapy ( FOLFIRI regimen, FOLFOX regimen or LV5FU2 regimen) + bevacizumab
- Chemotherapy (Active Comparator): Chemotherapy (FOLFIRI, FOLFOX, LV5FU2)
  Interventions: Drug: Chemotherapy ( FOLFIRI regimen, FOLFOX regimen or LV5FU2 regimen)

INTERVENTIONS:
Drug: Chemotherapy ( FOLFIRI regimen, FOLFOX regimen or LV5FU2 regimen)
  Arms: Chemotherapy
Drug: Chemotherapy ( FOLFIRI regimen, FOLFOX regimen or LV5FU2 regimen) + bevacizumab
  Arms: Chemotherapy associated with bevacizumab

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, irinotecan hydrochloride, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving bevacizumab together with combination chemotherapy may be a better way to block tumor growth. It is not yet known whether combination chemotherapy is more effective when given together with or without bevacizumab in treating patients with colorectal cancer.

PURPOSE: This randomized phase II trial is studying the side effects of giving bevacizumab together with first-line chemotherapy and to see how well it works in treating older patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate composite efficacy and safety, in terms of objective response or tumoral stability by RECIST criteria and no deterioration in the Spitzer QoL Index score of ≥ 2 points at 4 months, in older patients with unresectable metastatic colorectal adenocarcinoma treated with bevacizumab and first-line chemotherapy.
* To evaluate tolerance, in terms of no grade 4 arterial hypertension, grade 3-4 thromboembolic event, grade 3-4 cardiac insufficiency, and hospitalization not linked to chemotherapy, in these patients.

Secondary

* To evaluate toxicity in these patients.
* To assess time to deterioration of autonomy in these patients.
* To assess survival with no deterioration of autonomy of these patients.
* To evaluate time to deterioration of quality of life of these patients.
* To evaluate percentage of patients who received at least 2/3 of the protocol treatment at month 4.
* To assess time to treatment failure in these patients.
* To assess progression-free survival and global survival of these patients.

Tertiary

* To test for predictive factors of treatment success identified during the geriatric evaluation, according to the main judgment criterion, and analysis of the evolution of geriatric parameters during follow-up int these patients. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to chemotherapy (monotherapy vs double chemotherapy), primary tumor (resected vs non-resected), and quality-of-life score evaluated by the Spitzer QoL Index (0-3 vs 4-7 vs 8-10). Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive 1 of the following regimens according to the discretion of the investigator:

  * Simplified LV5FU2 comprising leucovorin calcium IV over 2 hours on days 1 and 15 and fluorouracil IV over 46 hours beginning on days 1 and 15.
  * FOLFIRI comprising leucovorin calcium IV over 2 hours on days 1 and 15; irinotecan hydrochloride IV over 2 hours on days 1 and 15; and fluorouracil IV over 46 hours beginning on days 1 and 15.
  * FOLFOX4 comprising oxaliplatin IV over 2 hours on days 1 and 15; leucovorin calcium IV over 2 hours on days 1 and 15; and fluorouracil IV over 46 hours beginning on days 1 and 15.

All treatment regimens repeat every 4 weeks for at least 6 months in the absence of disease progression or unacceptable toxicity.

* Arm B: Patients receive chemotherapy as in arm A. Patients also receive bevacizumab IV over 90 minutes on days 1 and 15. Treatment repeats every 4 weeks for at least 6 months in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed periodically. Blood specimens are collected for evaluation of the quantification of circulating cells for early prediction of response to treatment.

After completion of study therapy, patients are followed up every 2-3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic colorectal adenocarcinoma

  * Unresectable disease
* Measurable disease by RECIST criteria
* No cerebral metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Polynuclear neutrophils > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Proteinuria ≤ 1 g on 24-hour urine collection
* No unresolved intestinal occlusion or subocclusion
* No other progressive or unstabilized malignant tumor within the past 2 years
* No progressive gastroduodenal ulcer, wound, or bone fracture
* No active cardiac disease including any of the following:

  * Hypertension not adequately controlled
  * Myocardial infarction within the past 6 months
  * Poorly controlled angina
  * Decompensated congestive cardiac insufficiency
* No history of arterial thromboembolism or any of the following within the past 12 months:

  * Cerebrovascular accident
  * Transient ischemic attack
  * Subarachnoid hemorrhage
* No history of distal or visceral ischemic arterial pathology ≥ grade 2 within the past 12 months
* No history of life-threatening pulmonary embolism within the past 6 months
* Must have completed the geriatric self-administered questionnaire and the geriatric "team" questionnaire (including the Spitzer QoL Index)

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease

  * More than 6 months since adjuvant chemotherapy after resection of the primary tumor
* More than 4 weeks since major surgery, excluding biopsy
* More than 4 weeks since radiotherapy

Ages: 75 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Efficacy, in terms of objective response or tumoral stability by RECIST criteria | 4 months
Deterioration in the Spitzer QoL Index score of ≥ 2 points at baseline and at 4 months | 4 months
Tolerance, in terms of no grade 4 arterial hypertension, grade 3-4 thromboembolic event, grade 3-4 cardiac insufficiency, and hospitalization not related to chemotherapy | 4 months

SECONDARY OUTCOMES:
Toxicity | 4 months
Time to deterioration of autonomy | 4 months
Survival with no deterioration of autonomy | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aparicio, Principal Investigator — Hopital Avicenne
Locations (1):
- Hôpital Avicenne, Bobigny, France

REFERENCES:
- [Result] Aparicio T, Bouche O, Taieb J, Maillard E, Kirscher S, Etienne PL, Faroux R, Khemissa Akouz F, El Hajbi F, Locher C, Rinaldi Y, Lecomte T, Lavau-Denes S, Baconnier M, Oden-Gangloff A, Genet D, Paillaud E, Retornaz F, Francois E, Bedenne L; for PRODIGE 20 Investigators. Bevacizumab+chemotherapy versus chemotherapy alone in elderly patients with untreated metastatic colorectal cancer: a randomized phase II trial-PRODIGE 20 study results. Ann Oncol. 2018 Nov 1;29(11):2270. doi: 10.1093/annonc/mdx808. No abstract available. PMID 29718089